CLINICAL TRIAL: NCT03311516
Title: Evaluation of Insulin Therapy by Multiwave Bolus Based on the Lipid and Protein Content in Addition to the Carbohydrates Content Compared to Insulin Therapy Based Only on the Carbohydrates Content in type1 Diabetes Treated by Insulin Pump
Brief Title: New Insulin Therapy by Multiwave Bolus
Acronym: EVANEWFIT2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Central Hospital, Reims, France (Unknown); Central Hospital, Toulouse, France (Unknown); Central Hospital, Strasbourg, France (Unknown); Central Hospital, Besançon, France (Unknown); Central Hospital, Dijon, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A02414-49
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Type1diabetes
Keywords: insulin therapy
MeSH Terms: interventions — Lipids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A = intervention group (new functional insulin therapy) who adjusts the insulin bolus according to a dose titration algorithm taking into account the lipid and protein content in addition to that of carbohydrates. The functional insulin therapy is based on a Carbohydrate / Lipid / Protein count
  Interventions: Other: New functional insulin therapy
- Group B (Other): Group B=control group (functional insulin tehrapy) who adjusts the insulin bolus taking into account only the carbohydrate content. The functional insulin therapy is based on a Carbohydrate count only.
  Interventions: Other: functional insulin therapy

INTERVENTIONS:
Other: New functional insulin therapy — the patient receives the dietary devices and the instructions for the adaptation of the insulin bolus dose according to a new FIT
  Other Names: FIT based on a Carbohydrate / Lipid / Protein count
  Arms: Group A
Other: functional insulin therapy — the patient receives the dietary devices and the instructions for the adaptation of the insulin bolus dose according to FIT
  Other Names: FIT based on a carbohydrate count only
  Arms: Group B

SUMMARY:
The aim of the study is to evaluate the effect of insulin therapy when the bolus dose of insulin is calculated on the basis of protein and fat content in food intake, in addition to that of carbohydrates in T1D patients treated by insulin pump. The study is planned to recruit 150 patients with type1 diabetes already practicing functional insulin therapy based on carbohydrate counting in meals. We will therefore study the effect on continuous glucose measured by subcutaneous sensor, of meal bolus adjustments by comparing two groups of T1D patients:

* Groupe A takes into account the lipid and protein content in addition to the carbohydrate content
* Group B takes into account the carbohydrate content only At randomization, all patients receive dietary and adjustment of bolus doses instructions according to the randomization group. They have to apply these instructions for 3 months. At the end of 3 months, the study groups will be under glucose monitoring during two weeks in the Outpatient Clinic but returns to the investigational site in hospital to download data from the continuous measurement of glucose. In addition, we propose a period of extension similar to that of the main period, namely 3 months of application of dietetic and adaptation of bolus doses instructions and 2 weeks of continuous measurement of glucose.

During each 2 weeks period will be assessed specific glucose parameters in the post-prandial period over 4hours (glycemic sensor values in the glucose range between 70-140 mg / dl, glycemic sensor values in the glucose range between 140 -180 mg /dl and > 180 mg /dl) after taking each meal during the 13 days of Glucose Continuous Measurement (GCM), average daily glucose per meal, average blood glucose over the 13-day period after each meal.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic patient for more than one year, practicing functional insulin for at least 3 months but not more than 5 years
* Patient treated with external insulin pump (Medtronic or Omnipod pump)
* Patient performing intermittent blood glucose monitoring by the continuous interstitial glucose measurement system (Freestyle Libre) and who regularly wears this device with an achievement of at least 4 scans per day to obtain at least 90% of the possible values
* Patient with HbA1c ≤10.0% less than 3 months
* Patient with a willingness and ability to comply with study requirements and schedule of visits
* Patient who received complete information and signed informed consent

Exclusion Criteria:

* Patient with contraindication for rapid or ultra-rapid insulin analogues
* Patient for whom a change of insulin in the next 3 to 6 months is planned
* Women of childbearing age who do not have effective contraception
* Women who are pregnant or breast feeding or plan on becoming pregnant during the study
* Patient taking medication that interferes with interpretation of study results such as chronic corticosteroid therapy
* Patient with a chimio - or radiotherapy is in progress or is planned
* Patient abusing substances
* Patient who participated in another clinical study in the four weeks prior to inclusion
* Patient with or suspected of having any physical, psychological or cognitive disorders interfering with adherence to insulin therapy by pump, or compliance with dietary advice, or completion of the patient's diary
* Patient unable to comply with clinical guidelines, and unable to comply with 3-month follow-up
* Patient unable to understand information, to sign informed consent or to manage glycemic sensor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
The ratio of normoglycemia values to total glucose values | at 14 weeks since the patient randomization
  The ratio (expressed as a%) of the number of normoglycemia values over the total number of values collected over the 13-day period of the glucose monitoring

SECONDARY OUTCOMES:
Continuous Glucose Measurement (CGM) | at 14 weeks and at 28 weeks since the patient randomization
  Specific glycemic parameters in the post-prandial period over 4h (glycemic sensor values in the blood glucose range between 70-140 mg / dl, glycemic sensor values in the blood glucose area between 140 - 180 mg / dL and> 180 Mg / dl) after taking each meal during the 13 days of CGM, average daily glucose per meal, average blood glucose over the 13-day period after each meal
HbA1c | at 14 weeks and at 28 weeks since the patient randomization
  HbA1C dosage to assess glycemic control
Sensor wearing time | 12 weeks, 14 weeks, 26 weeks and 28 weeks since the patient randomization
  Sensor wearing time over the 3-month period and the 13-day CGM recording period
Number of sensor scans | 14 weeks and 28 weeks since the patient randomization
  Number of sensor scans performed by the patient with corresponding time periods
Number of boluses performed | at 14 weeks and at 28 weeks since the patient randomization
  Number of boluses performed over the 13-day period of the CGM
Satisfaction of the patient with regard to his treatment | at inclusion, at 12 weeks and 26 weeks since randomisation
  Patient satisfaction assessed by the DTSQs (status) and DTSQc (change)
Usability of the insulin pump | 14 weeks and 28 weeks since the patient randomization
  Evaluate the use of pump functions by patient ex. Bolus calculator, Temporary base rate

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Service d'Endocrinologie-Métabolisme et Diabétologie-Nutrition, Besançon
  - Service d'endocrinologie et maladies métaboliques, Dijon
  - Service d'Endocrinologie, Diabétologie et Nutrition, Nancy
  - Service Endocrinologie Diabète Nutrition, Reims
  - Structure d'Endocrinologie, Diabète et Nutrition, Strasbourg
  - Service de diabétologie, maladies métaboliques et nutrition, Toulouse